CLINICAL TRIAL: NCT00876486
Title: A Open-label, Randomized, Parallel, Phase III Trial to Evaluate the Efficacy and Safety of Genexol®-PM Compared to Genexol®(Conventional Paclitaxel With Cremorphor EL) in Subjects With Recurrent or Metastatic Breast Cancer
Brief Title: Evaluate the Efficacy and Safety of Genexol®-PM Compared to Genexol® in Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPMBC301
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genexol®-PM (Experimental): This is a open-labeled, randomized, parallel, phase III Trial. Up to 106 elgible patients will be enrolled in each treatment arm(Total 212 subjects will recruited) according to the trial design. Patients will be randomly allocated to arm A (Genexol-PM) or arm B (Paclitaxel).
  Interventions: Drug: Genexol-PM®
- Genexol® (Active Comparator): This is a open-labeled, randomized, parallel, phase III Trial. Up to 106 elgible patients will be enrolled in each treatment arm(Total 212 subjects will recruited) according to the trial design. Patients will be randomly allocated to arm A (Genexol-PM) or arm B (Paclitaxel).
  Interventions: Drug: Genexol®

INTERVENTIONS:
Drug: Genexol-PM® — Genexol-PM® 260mg/m2, intravenous infusion over 3 hours, every 3 weeks
  Arms: Genexol®-PM
Drug: Genexol® — Genexol® 175mg/m2, intravenous infusion over 3 hours, every 3 weeks
  Arms: Genexol®

SUMMARY:
Phase III trial to evaluate the efficacy and safety of Genexol®-PM compared to Genexol® in subjects with recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects should meet all of the following criteria to participate in the trial.

1. Subjects who aged 18 years or older.
2. Subjects whose written informed consent was obtained complying with the local regulatory requirements prior to their participation in the trial.
3. Subjects who have histologically or cytologically confirmed breast cancer with evidence of recurrence or metastasis.
4. If subjects have received Taxanes as neo-adjuvant or adjuvant therapy, the subjects should have relapsed with breast cancer after 12 months of completing neo-adjuvant or adjuvant therapy with Taxanes.
5. Subjects who have measurable disease in accordance with the RECIST criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  Evaluate the efficacy of Genexol®-PM versus Genexol® in subjects with recurrent or metastatic breast cancer based on Objective Response Rate.

SECONDARY OUTCOMES:
Overall Survival, Progress Free Survival, Time to Tumor Progression, Duration of Overall Response | Event driven
  To evaluate the efficacy of Genexol®-PM relative to Genexol® as measured by Overall Survival, Progress Free Survival, Time to Tumor Progression, Duration of Overall Response.
Safety and toxicity | Throughout study
  To compare the safety and toxicity of Genexol®-PM with those of Genexol®

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea